CLINICAL TRIAL: NCT00218725
Title: Cognitive Therapy for Suicide Attempters With Drug Dependence Disorder
Brief Title: Effectiveness of Cognitive Therapy for Suicide Attempters With Drug Dependence Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20MH071905-02 (NIH); P20MH071905-02 (NIH); 802439 (Other: University of Pennsylvania IRB); FWA00003616; DSIR 83-ATP
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Suicide, Attempted; Substance-Related Disorders
Keywords: Cognitive Therapy; Suicide; Addictions; Substance Abuse
MeSH Terms: conditions — Suicide, Attempted; Substance-Related Disorders; Suicide; Behavior, Addictive | interventions — Cognitive Behavioral Therapy; Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Therapy (Other): The cognitive therapy intervention for suicide attempters has been designed to provide a brief, timely, flexible intervention that can be incorporated into general and psychiatric inpatient and outpatient services and applied to the population of patients who attempt suicide. A central feature of the intervention is the adaptation of cognitive therapy to the population of patients who attempt suicide. The focus of the intervention is the identification of core beliefs and key automatic thoughts that were elicited prior to and during the most recent suicide attempt. Once these beliefs and thoughts have been articulated, the counselor and patient develop more adaptive responses during an acute suicidal crisis.
  Interventions: Behavioral: Cognitive Therapy
- Enriched Care (Other): The Enriched Care condition will be used as the treatment comparison condition for this study. The Enriched Care condition consists of the usual care that patients may obtain in the community as well as the assessment and referral services provided by the case managers. Participation in the study does not restrict patients in any way in their access to other health care, and all patients in both conditions will be allowed to receive any additional mental health and substance abuse treatment in the community.
  Interventions: Other: Enriched Care

INTERVENTIONS:
Behavioral: Cognitive Therapy — The cognitive therapy intervention for suicide attempters has been designed to provide a brief, timely, flexible intervention that can be incorporated into general and psychiatric inpatient and outpatient services and applied to the population of patients who attempt suicide. A central feature of the intervention is the adaptation of cognitive therapy to the population of patients who attempt suicide. The focus of the intervention is the identification of core beliefs and key automatic thoughts that were elicited prior to and during the most recent suicide attempt. Once these beliefs and thoughts have been articulated, the counselor and patient develop more adaptive responses during an acute suicidal crisis.
  Arms: Cognitive Therapy
Other: Enriched Care — The Enriched Care condition will be used as the treatment comparison condition for this study. The Enriched Care condition consists of the usual care that patients may obtain in the community as well as the assessment and referral services provided by the case managers. Participation in the study does not restrict patients in any way in their access to other health care, and all patients in both conditions will be allowed to receive any additional mental health and substance abuse treatment in the community.
  Other Names: Case Management
  Arms: Enriched Care

SUMMARY:
This study will examine the effectiveness of combining cognitive therapy with enriched usual care for preventing subsequent suicide attempts in people with a drug dependence who have recently attempted suicide.

DETAILED DESCRIPTION:
Suicide attempts involving drug abuse are a major public health problem. Development of interventions that focus on reducing the suicide attempt rate among drug abusers is a necessity. There is a strong connection between drug abuse and both suicide attempts and completed suicide. As much as 45% of drug abusers have attempted suicide at least once. The rate of completed suicide among drug abusers has been reported to be as much as 30 times the rate for the general population. Unfortunately, there is a lack of empirically supported treatments for reducing suicidal behavior in drug abusers. This study will develop and evaluate the effectiveness of a cognitive therapy intervention for people with a drug dependence disorder who recently attempted suicide.

Participants in this single-blind study will be randomly assigned to one of two treatment groups: cognitive therapy combined with enriched usual care; or enriched usual care alone. An initial baseline assessment will occur within 7 days following the participant's suicide attempt and subsequent medical evaluation at a hospital emergency department. Suicide behavior and ideation, depression, hopelessness, and addiction severity will be assessed. Following the baseline assessment, treatment will begin. The cognitive therapy treatment will be specifically developed to prevent suicide attempts. It will involve the identification of proximal thoughts, images, and core beliefs that were activated prior to the suicide attempt. Cognitive and behavioral strategies will be applied to address the identified thoughts and beliefs. Patients will also learn adaptive ways of coping with stressors. The enriched usual care will entail standard treatments for suicide prevention. Study visits will occur 1, 3, 6, 12, 18, and 24 months following enrollment. Baseline measurements will be repeated at each study visit to evaluate participants' improvement. Participants receiving cognitive therapy will attend approximately 10 weekly or bi-weekly outpatient study visits. Participation will last for 2 years.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00149773

ELIGIBILITY:
Inclusion Criteria:

* Recent suicide attempt with an emergency department visit within 48 hours of the attempt (suicide attempt is considered to be a potentially self-injurious behavior with a nonfatal outcome for which there is evidence, either explicit or implicit, that the individual intended to kill himself or herself)
* Current DSM-IV diagnosis of a current drug dependence disorder within the past 6 months

Exclusion Criteria:

* Self-mutilating behavior without intent to commit suicide
* An acute, unstable, or severe Axis III disorder that may affect participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Suicidal Attempts | Months 1, 3, 6, 12, 18, and 24

SECONDARY OUTCOMES:
Suicide Ideation | Months 1, 3, 6, 12, 18, and 24
Depression | Months 1, 3, 6, 12, 18, and 24
Hopelessness | Months 1, 3, 6, 12, 18, and 24
Substance Use | Months 1, 3, 6, 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T. Beck, MD, Principal Investigator — University of Pennsylvania; Gregory K. Brown, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Psychopathology Research Unit-University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617